Pain Outcomes of Intra-operative IV Tylenol and/or Toradol for Carpal Tunnel and Distal Radius Fracture Surgeries

NCT 02313675

Initial IRB approval: 5/11/15 Most recent IRB renewal: 1/25/17 An a priori power analysis determined that eleven subjects per treatment group were required (total of 44 patients) to detect a difference in the 11-point pain score of 1.0 between groups. Patients recorded pain levels at 8 hour intervals and daily opioid use for seven days after surgery. Data analysis included calculation of descriptive statistics including frequency counts and percentages for categorical variables and measures of central tendency (means, medians) and dispersion (standard deviations, ranges) for continuous variables. ANOVA and Kruskal-Wallis tests were used to compare mean pain and opioid consumption between groups.